CLINICAL TRIAL: NCT06578676
Title: A Clinical Study to Evaluate the Safety and Pharmacokinetic Interaction Between HODO-22251 and HODO-22252 in Healthy Adults
Brief Title: To Evaluate the Safety and Pharmacokinetic Interaction Between HODO-22251 and HODO-22252 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HD-EZE-01
Record Dates: First submitted 2024-07-04; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Dyslipidemias
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — empagliflozin; Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: 2 sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 25mg (Experimental): * Period 1: Empagliflozin (QD, 5d)
  * wash-out: 7d
  * Period 2: Ezetimibe/Rosuvastatin (QD, 2d) and Empagliflozin and Ezetimibe/Rosuvastatin (QD, 5d)
  Interventions: Drug: Empagliflozin 25 MG; Drug: Ezetimibe/Rosuvastatin 10/10mg; Drug: Empagliflozin 25 MG with Ezetimibe/Rosuvastatin 10/10mg
- Rosuvastatin/Ezetimibe 10/10mg (Experimental): * Period 1: Ezetimibe/Rosuvastatin (QD, 7d)
  * wash-out: 14d
  * Period 2: Ezetimibe/Rosuvastatin (QD, 2d) and Empagliflozin and Ezetimibe/Rosuvastatin (QD, 5d)
  Interventions: Drug: Ezetimibe/Rosuvastatin 10/10mg; Drug: Empagliflozin 25 MG with Ezetimibe/Rosuvastatin 10/10mg

INTERVENTIONS:
Drug: Empagliflozin 25 MG — PO, QD
  Arms: Empagliflozin 25mg
Drug: Ezetimibe/Rosuvastatin 10/10mg — PO, QD
Drug: Empagliflozin 25 MG with Ezetimibe/Rosuvastatin 10/10mg — PO, QD

SUMMARY:
The purpose of this study is to evaluate pharmacokinetic interaction and safety of co-administrated 25mg of Empagliflozin and 10/10mg Ezetimibe/Rosuvastatin in steady state in healthy volunteers.

DETAILED DESCRIPTION:
This trial is a phase 1 study to evaluate pharmacokinetic interaction and safety of co-administrated 25mg of Empagliflozin and 10/10mg of Ezetimibe/Rosuvastatin in steady state in healthy volunteers.

This is open-label, multiple-dose, two-arm, two-period and fixed-sequence design.

In Arm A, 18 subjects will be assigned. The subjects take 25mg of empagliflozin for 5days(Period 1). After 7days of washout period, the subjects take 10/10mg of Ezetimibe/Rosuvastatin for 2days and take co-administrated 25mg of Empagliflozin and 10/10mg of Ezetimibe/Rosuvastatin for 5days.

In Arm B, 38 subjects will be assigned. The subjects take 10/10mg of Ezetimibe/Rosuvastatin for 7days(Period 1). After 14days of washout period, the subjects take 25mg of empagliflozin for 2days and take co-administrated 25mg of Empagliflozin and 10/10mg of Ezetimibe/Rosuvastatin for 5days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age: 19 and over , healthy volunteer
* Body mass index (BMI): 18.5≤BMI≤29.9 kg/m²

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination or effects of the study drugs will not be normal
* Clinically relevant findings(e.g. blood pressure, electrocardiogram(ECG); physical and gynecological examination, laboratory examination)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of Empagliflozin, Total Ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48hours of after administration
  Cmax,ss of Empagliflozin, Total Ezetimibe and Rosuvastatin
AUCtau,ss of Empagliflozin, Total Ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  AUCtau,ss of Empagliflozin, Total Ezetimibe and Rosuvastatin

SECONDARY OUTCOMES:
Vdss/F of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  Vdss/F of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
Cmax,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  Cmax,ss, AUCtau,ss, AUCinf,ss, Tmax,ss, Cmin,ss, t1/2,ss, CLss/F, Vdss/F of Free ezetimibe
AUCtau,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  AUCtau,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
AUCinf,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  AUCinf,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
Tmax,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  Tmax,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
Cmin,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  Cmin,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
t1/2,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  t1/2,ss of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin
CLss/F of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72hours of after administration
  CLss/F of Free ezetimibe, Empagliflozin, Total ezetimibe and Rosuvastatin

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university hospital, Daegu, Gyeongsangbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No